CLINICAL TRIAL: NCT05867589
Title: Study of Novel PET Tracer Gallium [68Ga]/ Fluorine [18F] -FAPI-04 in the Diagnosis of Cardiovascular Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, FengWang, Director of nuclear medicine department, Nanjing First Hospital, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20230428-02
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Myocardial Fibrosis
Keywords: Fibroblast Activation Protein, PET-MRI,myocardial fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga/18F-FAPI-04 (Experimental): For the injection, subjects will receive a target dose of 0.1~0.15mCi/Kg 68Ga/18F-FAPI-04 as a bolus injection.
  Interventions: Drug: 68Ga/18F-FAPI-04

INTERVENTIONS:
Drug: 68Ga/18F-FAPI-04 — Subjects will receive one injection of 68Ga/18F-FAPI-04 (0.1~0.15mCi/Kg), a PET radiopharmaceutical selective for fibroblast activation protein. 68Ga/18F-FAPI-04 injection will be followed by a 10 ml saline flush.

SUMMARY:
The purpose of this study is to evaluate the safety of fibroblast activating protein receptor imaging agent [68Ga]/ Fluorine [18F] -fibroblast activating protein inhibitor (68Ga/18F-FAPI-04) in clinical application and to verify its effectiveness in the diagnosis of cardiovascular diseases.

DETAILED DESCRIPTION:
The implementation of this project will promote the research of PET-MRI molecular imaging using the new nuclide imaging with the target of FAP combined with the MRI T1 mapping and ECV measurement technology, realize the fusion of nuclear medicine and magnetic resonance technology in a real sense, dynamically monitor the occurrence and development of myocardial fibrosis in heart failure at an early stage, and establish a complete set of myocardial fibrosis imaging programs. To provide an important basis for the exploration of anti-fibrosis therapy in heart failure and accelerate the pace of clinical transformation of this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary subjects, patients or their legal representatives to sign informed consent;
2. There was no limitation on the gender of the volunteers, whose age ranged from 18 to 85 years old, including the cut-off value;
3. Myocardial injury caused by various causes was found by other imaging methods (cardiac ultrasound, coronary angiography, coronary CT, cardiac MRI, etc.);
4. Kidney GFR > 50 ml/min, ERPF > 280 ml/min, platelet count (PLT) > 75 000/μL, leukocyte (WBC) > 3000/μL, alanine aminotransferase ALT, aspartate aminotransferase AST < 3 times the normal value.

Exclusion Criteria:

1. Allergic to the same drugs (drugs with similar chemical or biological components to fibroblast activating protein inhibitors), allergic constitution or currently suffering from allergic diseases;
2. Clinical investigators who are currently conducting clinical studies on other drugs, or who have participated in any drug (excluding vitamins and minerals);
3. Have other clinical problems that are difficult to control (such as HIV, hepatitis C virus infection or active hepatitis B, or other severe chronic infections and serious mental, neurological, respiratory and other diseases);
4. Red blood cell RBC is less than 4×1012, white blood cell WBC is less than 3×109, hemoglobin is less than 80g/L, PLT is less than 75,000 ×109;
5. Significantly abnormal liver and kidney function, GFR less than 20 ml/min;
6. Cardiac ejection fraction (EF) was assessed to be less than 10%;
7. The expected survival time is less than half a year; Coronary stent implantation within 2 weeks or coronary artery bypass graft within 6 months;
8. Severe acute concomitant disease or severe refractory mental disorder;
9. Pregnant and lactating women (pregnancy is defined as positive in blood pregnancy studies);
10. Patients whose physical conditions are not suitable for radioactive examination;
11. Patients with metal implants (pacemakers, etc.) or spatial claustrophobia or other MRI related contraindications;
12. Any situation that the presiding officer of this study believes may cause harm or potential harm to any link related to this test.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of 68Ga/18F-FAPI-04 Uptake Patterns by Regional SUV Values | 31 months
  68Ga/18F-FAPI-04 uptake patterns will be assessed in regions of interest (ROIs) which relevant to myocardial fibrosis pathology. Standard uptake value (SUV) will be calculated for each ROI, and standardized uptake value ratios (SUVRs) will be calculated by normalizing SUV of ROIs to the SUV of relevant reference region.
Safety and Tolerability Profile Measured by Adverse Events (AEs) | 31 months
  Safety and tolerability profile for the administration of 68Ga/18F-FAPI-04 and positron emission tomography (PET) scanning are measured by number of participants with adverse events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Study Director — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Luo R, Zhao Z, Zhang C, Li RS, Wang Y, Meng Q, Ni Y, Wang B, Li L, Feng L, Yang R, Xie L, Chen X, Zhang MR, Wang F. Evaluation of myocardial fibrosis and wall motion abnormality with 68Ga-FAPI PET/MR in coronary heart disease. EJNMMI Res. 2025 Jul 21;15(1):89. doi: 10.1186/s13550-025-01246-2. PMID 40690085